CLINICAL TRIAL: NCT05052502
Title: Targeting High-risk Populations With Enhanced Reactive Focal Mass Drug Administration: A Study to Assess the Effectiveness and Feasibility for Plasmodium Falciparum and Plasmodium Vivax Malaria in Thailand
Brief Title: Targeting High Risk Populations With Enhanced Reactive Focal Mass Drug Administration in Thailand
Acronym: COMBAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: Center for Malariology, Parasitology, and Entomology (Unknown); Tulane University School of Public Health and Tropical Medicine (Other); University of Massachusetts, Amherst (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 19-04062020
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Plasmodium Falciparum Malaria; Plasmodium Vivax Malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- reactive focal mass drug administration (rfMDA) (Experimental): Reactive FMDA (rfMDA) led by VMVs in response to cases in study area sub-district, in both villages and forest workers; quantitative G6PD testing for all individuals and 14-day PQ for G6PD non-deficient.
  Interventions: Other: Case Management and Follow-up; Other: Reactive focal mass drug administration (rfMDA)
- Control (Active Comparator): Standard of care including case management through health facilities and malaria posts/VMVs; village-based RACD conducted by district staff in some areas.
  Interventions: Other: Case Management and Follow-up

INTERVENTIONS:
Other: Case Management and Follow-up — Individuals will be told of their test result and a positive test result on either RDT will prompt treatment as per the national treatment guidelines.
  * Individuals with P. falciparum infection will be treated with an age-appropriate course of dihydroartemisinin/piperaquine (DHAP) or artesunate-pyronaridine (Pyramax) and PQ.
  * At all study sites in Thailand, patients with a P. vivax infection identified by the standard combination RDT will be tested by the VMV and Health Promotion Hospital (HPH) staff member using the quantitative G6PD RDT. G6PD normal individuals will be treated with Chloroquine (CQ) and a 14-day course of primaquine (PQ). G6PD deficient individuals will receive CQ alone and referred to the nearest health facility for further primaquine management decisions.
Other: Reactive focal mass drug administration (rfMDA) — Reactive focal mass administration (rfMDA) will be implemented around the index case household and to forest co-workers/co-travelers in Thailand. The VMV will conduct the investigation visit within 7 days after the notification of the index case. All members of the index case's household as well as all members of the nearest five households around the index case's household, including temporary visitors will be invited to participate in the study and to be treated for malaria without a malaria test. After obtaining participants' or parents/guardians' consent, the VMV will proceed with the participant questionnaire, and all consenting household members will be tested for G6PD using the G6PD quantitative test prior to administration of antimalarials.
  For rfMDA, all eligible participants will be offered artesunate-mefloquine (AS-MQ). Per national policy, a 14-day course of primaquine will be administered to G6PD non-deficient study participants.
  Arms: reactive focal mass drug administration (rfMDA)

SUMMARY:
This study assesses the effectiveness of reactive focal mass drug administration (rfMDA), targeting both village and forest working populations, compared to control for reducing the health promotion hospital-level (sub-district) incidence and prevalence of P. falciparum and P. vivax within five provinces in Thailand.

DETAILED DESCRIPTION:
Thailand currently has a well-developed and robust surveillance system based on detailed mapping of all cases to the village foci level and stratification of response. In fiscal year 2019, 5,833 cases of malaria were reported with 83.0% P. vivax and 12.9% P. falciparum; nine deaths were reported. This represents a 20.8% decrease in total cases from fiscal year 2018. Currently, there are 701 "A1" villages in 44 provinces.

The research proposed here will evaluate the effectiveness and feasibility of enhanced reactive focal mass drug administration, results of which will have direct implications for continued roll out the community-led foci management, providing practical guidance that other malaria programs can utilize. Responding to the malaria among high risk populations is a requirement from the National Malaria Elimination Strategy in Thailand. Additionally, Thailand has experienced outbreaks related to forest work over the past several years, and consequently the Department of Vector Borne Disease (DVBD) is interested in introducing more aggressive parasite elimination strategies, including rfMDA for P. falciparum and P. vivax specifically targeting high-risk populations to interrupt transmission and rapidly accelerate elimination.

ELIGIBILITY:
Inclusion Criteria for rfMDA:

* Index cases: Presented as a confirmed malaria case to an intervention health facility or village malaria worker, and lives in a village within a selected intervention subdistrict, or worked or spent at least one night at a forest or forest-fringe site in the past 30 days located within an intervention subdistrict
* Village residents: Lives in a village within a selected intervention subdistrict area and in one of the five households closest to the residence of an index case of malaria
* Co-worker/traveler referral: Worked or traveled and spent at least one night in forest in past 30 days in same location within an intervention subdistrict as an index case of malaria
* All participants: Willing and available to participate in the study and informed consent for participant under the age of 18 will be provided by the parent or guardian. Participants for focus group discussions (FGDs) and key informant interviews (KIIs); 18 years of age or older

Exclusion Criteria:

• For rfMDA:

* Previous participation in the study as a result of any rfMDA event in the past 30 days
* Individuals with severe disease or drug contra-indications will be excluded from the treatment component only
* Artesunate-Mefloquine: Pregnancy in the first trimester, or known drug allergy
* Use of Mefloquine within 60 days of first treatment prior to enrollment date.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49118 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed P. falciparum and P. vivax malaria parasite incidence | 3 months
  Defined as the number of outpatient (OPD) malaria confirmed and suspected cases per person per year for each sub-district, as ascertained from the health facility registers, utilizing administrative catchment population size estimates for the exposure denominator.
PCR-based P. falciparum and P. vivax parasite prevalence in sampled sub-districts | 3 months
  Defined as the proportion of individuals ≥18 months old with P. falciparum or P. vivax infection (detected by PCR) out of all individuals ≥18 months tested within the end line survey.

SECONDARY OUTCOMES:
Population coverage of rfMDA interventions | 3 months
  This indicator will be measured in two ways. Operational program coverage will be defined as the proportion of individuals ≥18 months old and households visited and offered the rfMDA interventions within the target areas per time period. Effective program coverage is defined as the proportion of individuals (≥18 months old) that agreed to participate in the rfMDA intervention among all individuals ≥18 months old eligible to participate in the intervention in the target population per time period.
Feasibility of conducting rfMDA at the community level | 3 months
  Feasibility will be determined based upon a combination of population coverage data, responses of provincial, district, and health staff, VMWs, and community members to interviews and focus groups at baseline and end line, village malaria workers (VMWs) competency checklists at baseline, midline, and end line, and cost data.
Acceptability of rfMDA approach | 3 months
  Acceptability will be determined based upon refusal rates during interventions and responses of community members and VMWs to end line questionnaire, interviews, and focus groups.
Adverse event rate | 3 months
  Safety measures will include the adverse event rate amongst treated individuals and hemoglobin measurement pre and post treatment for individuals receiving PQ.
Operational feasibility of glucose-6-phosphate dehydrogenase (G6PD) testing and referral | 3 months
  Operational feasibility of G6PD testing and referral will be determined by responses of health staff and VMWs to interviews and focus groups at baseline and end line and competency checklists at baseline, midline, and end line, the proportion of P. vivax cases with a valid G6PD result, and proportion of referred cases presenting at a health facility for G6PD testing.
Assessment of P. vivax treatment adherence | 3 months
  Treatment adherence will be determined by the proportion of P. vivax cases with physical evidence of adherence through pill count and the P. vivax relapse rate across study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bennett, MA, PhD, Principal Investigator — University of California, San Francisco; Cheewanan Lertpiriyasuwat, MD, Principal Investigator — Ministry of Health, Thailand
Locations (1):
- Division of Vector Born Diseases, Ministry of Health, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any parties outside of the study team.

REFERENCES:
- [Background] Bousema T, Griffin JT, Sauerwein RW, Smith DL, Churcher TS, Takken W, Ghani A, Drakeley C, Gosling R. Hitting hotspots: spatial targeting of malaria for control and elimination. PLoS Med. 2012 Jan;9(1):e1001165. doi: 10.1371/journal.pmed.1001165. Epub 2012 Jan 31. PMID 22303287
- [Background] Cotter C, Sturrock HJ, Hsiang MS, Liu J, Phillips AA, Hwang J, Gueye CS, Fullman N, Gosling RD, Feachem RG. The changing epidemiology of malaria elimination: new strategies for new challenges. Lancet. 2013 Sep 7;382(9895):900-11. doi: 10.1016/S0140-6736(13)60310-4. Epub 2013 Apr 15. PMID 23594387
- [Background] Moonen B, Cohen JM, Snow RW, Slutsker L, Drakeley C, Smith DL, Abeyasinghe RR, Rodriguez MH, Maharaj R, Tanner M, Targett G. Operational strategies to achieve and maintain malaria elimination. Lancet. 2010 Nov 6;376(9752):1592-603. doi: 10.1016/S0140-6736(10)61269-X. Epub 2010 Oct 28. PMID 21035841
- [Background] Hustedt J, Canavati SE, Rang C, Ashton RA, Khim N, Berne L, Kim S, Sovannaroth S, Ly P, Menard D, Cox J, Meek S, Roca-Feltrer A. Reactive case-detection of malaria in Pailin Province, Western Cambodia: lessons from a year-long evaluation in a pre-elimination setting. Malar J. 2016 Mar 1;15:132. doi: 10.1186/s12936-016-1191-z. PMID 26931488
- [Background] Rossi G, Van den Bergh R, Nguon C, Debackere M, Vernaeve L, Khim N, Kim S, Menard D, De Smet M, Kindermans JM. Adapting Reactive Case Detection Strategies for falciparum Malaria in a Low-Transmission Area in Cambodia. Clin Infect Dis. 2018 Jan 6;66(2):296-298. doi: 10.1093/cid/cix781. PMID 29020325
- [Background] Das S, Peck RB, Barney R, Jang IK, Kahn M, Zhu M, Domingo GJ. Performance of an ultra-sensitive Plasmodium falciparum HRP2-based rapid diagnostic test with recombinant HRP2, culture parasites, and archived whole blood samples. Malar J. 2018 Mar 17;17(1):118. doi: 10.1186/s12936-018-2268-7. PMID 29549888
- [Background] World Health Organization. (2015). Guidelines for the treatment of malaria. World Health Organization
- [Background] Landier J, Parker DM, Thu AM, Lwin KM, Delmas G, Nosten FH; Malaria Elimination Task Force Group. Effect of generalised access to early diagnosis and treatment and targeted mass drug administration on Plasmodium falciparum malaria in Eastern Myanmar: an observational study of a regional elimination programme. Lancet. 2018 May 12;391(10133):1916-1926. doi: 10.1016/S0140-6736(18)30792-X. Epub 2018 Apr 24. PMID 29703425
- [Background] Howes RE, Dewi M, Piel FB, Monteiro WM, Battle KE, Messina JP, Sakuntabhai A, Satyagraha AW, Williams TN, Baird JK, Hay SI. Spatial distribution of G6PD deficiency variants across malaria-endemic regions. Malar J. 2013 Nov 15;12:418. doi: 10.1186/1475-2875-12-418. PMID 24228846
- [Background] White MT, Karl S, Battle KE, Hay SI, Mueller I, Ghani AC. Modelling the contribution of the hypnozoite reservoir to Plasmodium vivax transmission. Elife. 2014 Nov 18;3:e04692. doi: 10.7554/eLife.04692. PMID 25406065
- [Background] Douglas NM, Poespoprodjo JR, Patriani D, Malloy MJ, Kenangalem E, Sugiarto P, Simpson JA, Soenarto Y, Anstey NM, Price RN. Unsupervised primaquine for the treatment of Plasmodium vivax malaria relapses in southern Papua: A hospital-based cohort study. PLoS Med. 2017 Aug 29;14(8):e1002379. doi: 10.1371/journal.pmed.1002379. eCollection 2017 Aug. PMID 28850568
- [Background] Ministry of Health Lao PDR. The Evaluation of G6PD Rapid Tests and the Use of Primaquine for the Treatment of Plasmodium Vivax Infections in Luangprabang, Savannakhet and Champasak Provinces (Apr-Nov 2015). (2015)
- [Background] Center for Malariology Parasitology and Entomology Lao PDR. Lao PDR Malaria National Strategic Plan 2016-2020. (2015).
- [Background] WHO. Updated WHO policy recommendation: Single dose primaquine as a gametocytocide in Plasmodium falciparum malaria. World Health Organisation (2012).
- [Background] Baum E, Sattabongkot J, Sirichaisinthop J, Kiattibutr K, Davies DH, Jain A, Lo E, Lee MC, Randall AZ, Molina DM, Liang X, Cui L, Felgner PL, Yan G. Submicroscopic and asymptomatic Plasmodium falciparum and Plasmodium vivax infections are common in western Thailand - molecular and serological evidence. Malar J. 2015 Feb 25;14:95. doi: 10.1186/s12936-015-0611-9. PMID 25849211
- [Background] Corran P, Coleman P, Riley E, Drakeley C. Serology: a robust indicator of malaria transmission intensity? Trends Parasitol. 2007 Dec;23(12):575-82. doi: 10.1016/j.pt.2007.08.023. Epub 2007 Nov 7. PMID 17988945
- [Background] Chan CW, Sakihama N, Tachibana S, Idris ZM, Lum JK, Tanabe K, Kaneko A. Plasmodium vivax and Plasmodium falciparum at the crossroads of exchange among islands in Vanuatu: implications for malaria elimination strategies. PLoS One. 2015 Mar 20;10(3):e0119475. doi: 10.1371/journal.pone.0119475. eCollection 2015. PMID 25793260
- [Background] Beutler E, Duparc S; G6PD Deficiency Working Group. Glucose-6-phosphate dehydrogenase deficiency and antimalarial drug development. Am J Trop Med Hyg. 2007 Oct;77(4):779-89. PMID 17978087
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546